CLINICAL TRIAL: NCT04410432
Title: Immune Response and Risk of Serious Infection to SARS-Cov2
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GHESQUIERE AOIc 2020
Record Dates: First submitted 2020-05-29; First posted 2020-06-01 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: SARS Cov2, Immune Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient: Patient hospitalized with SARS-Cov2 infection proven by virological sampling.
  Interventions: Biological: Blood sample collection

INTERVENTIONS:
Biological: Blood sample collection — Additional blood volumes taken during a routine care blood test:
  * 1 dry tube 5 mL for isolation and freezing of serum
  * 1 x 5 mL EDTA tube to isolate and freeze plasma
  * 8 heparinized 6 mL tubes for flow cytometry study

SUMMARY:
To date, nearly 2 million people, including at least 100,000 in France, have been infected with SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2). This infection is very heterogeneous in nature, ranging from asymptomatic forms to acute respiratory distress syndrome patterns in 6.1% of cases, leading to an estimated overall mortality of 5.2%.

Apart from age, few risk factors for a pejorative evolution have been identified: arterial hypertension, diabetes, cardiovascular history, obesity and chronic respiratory pathology in particular. The median incubation period is 5 days and the median time between the appearance of the first symptoms and the onset of hypoxia requiring admission to intensive care is 7 to 12 days. The mechanisms involved in the occurrence of these secondary worsening patterns are unclear. One hypothesis is that it is related to an inappropriate inflammatory response rather than a direct cytopathic effect of the virus. The objective of this study is to measure the intensity of the T lymphocyte response in patients hospitalized for Cov2 SARS infection in order to determine whether the intensity of the response is associated with worsening of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Person having given his or her non-opposition
* Patient hospitalized with an SARS-Cov2 infection proven by virological sampling (nasopharyngeal or sputum PCR) less than 8 days old.

Exclusion Criteria:

* Person subject to a legal protection measure (curatorship, guardianship)
* Person subject to a safeguard measure of justice
* Pregnant, parturient or breastfeeding woman
* Major incapable or incapable of giving consent
* Minor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for SARS-Cov-2 infection
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Percentage of circulating Th1 lymphocytes | Until the end of the study, about 12 months.
  Flow cytometry measurement of the percentage of circulating Th1 lymphocytes

SECONDARY OUTCOMES:
Serum IFN concentrations-γ, CXCL9, CXCL10, CXCL11 | Until the end of the study, about 12 months.
  Immunofluorimetric measurement of serum concentrations of IFN-γ, CXCL9, CXCL10, CXCL11

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

REFERENCES:
- [Result] Samson M, Nicolas B, Ciudad M, Greigert H, Guilhem A, Cladiere C, Straub C, Blot M, Piroth L, Rogier T, Devilliers H, Manckoundia P, Ghesquiere T, Francois S, Lakomy D, Audia S, Bonnotte B. T-cell immune response predicts the risk of critical SARS-Cov2 infection in hospitalized COVID-19 patients. Eur J Intern Med. 2022 Aug;102:104-109. doi: 10.1016/j.ejim.2022.06.001. Epub 2022 Jun 3. PMID 35690570